CLINICAL TRIAL: NCT00314821
Title: A Randomized, Double-blind, Placebo-controlled Study of the Efficacy of Ropinirole in the Treatment of Depression in Bipolar Disorder
Brief Title: Ropinirole in the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Emory University (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHA-IRB-0116/05/05
Record Dates: First submitted 2006-04-13; First posted 2006-04-17 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder, ropinirole, depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — ropinirole

INTERVENTIONS:
Drug: ropinirole

SUMMARY:
To demonstrate efficacy and safety of Requip in in treating bipolar depression.

DETAILED DESCRIPTION:
This study is 8 weeks long, with an optional additional 8 weeks. The study is placebo-controlled and patients are randomized to receive either ropinerol or placebo. Changes in depression, anxiety and overall psychiatric symptoms will be monitored during participation.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for bipolar disorder
* Current MADRS score > 16
* Current MRS-SADS score < 10
* Prior to participation in this study, each subject must sign an informed consent.
* All patients will be required to also take at least one other mood-stabilizing agent, defined as a standard agent (lithium, valproate, carbamazepine) or a novel anticonvulsant agent (oxcarbazepine, gabapentin, topiramate). If patients are not taking any of these agents on study initiation, they will be required to start one of these agents at study initiation. Study inclusion criteria must be met after at least 2 weeks of treatment with one of these mood-stabilizing agents.

Exclusion Criteria:

* Any serious acute medical illness
* Any clinically serious evidence of suicidality or score of 3 or greater on suicide item on MADRS scale

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09 (Actual); Primary Completion 2007-06-01 (Actual); Study Completion 2008-03-17 (Actual)

PRIMARY OUTCOMES:
Primary outcome will be group differences between Requip and placebo in random effects linear regression analysis.

SECONDARY OUTCOMES:
The secondary outcomes will include predictors of response, such as insight into illness, comorbid anxiety symptoms, prior course of illness, previous treatment history with antidepressants, and other relevant clinical and demographic features.

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Dunn, MD,PhD, Principal Investigator — Cambridge Health Alliance
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - Cambridge Health Alliance, Cambridge, Massachusetts